CLINICAL TRIAL: NCT06425874
Title: The Impact of Socioeconomic Determinants on the Patient Reported Outcomes in Young Breast Cancer Patients After Breast Surgery: an Observational Cohort Study
Brief Title: The Impact of Socioeconomic Determinants on the Patient Reported Outcomes in Young Breast Cancer Patients After Breast Surgery
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Kai, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-147-01
Record Dates: First submitted 2024-04-29; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Surgery; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy; Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast-conserving surgery
  Interventions: Procedure: Breast-conserving surgery
- Mastectomy
  Interventions: Procedure: Mastectomy
- Mastectomy with reconstruction
  Interventions: Procedure: Mastectomy with reconstruction

INTERVENTIONS:
Procedure: Breast-conserving surgery — Breast-conserving surgery
  Groups: Breast-conserving surgery
Procedure: Mastectomy — Mastectomy without reconstruction
  Groups: Mastectomy
Procedure: Mastectomy with reconstruction — Any type of reconstruction(include implant and autologous)
  Groups: Mastectomy with reconstruction

SUMMARY:
Breast-conserving surgery is the standard treatment for young breast cancer patients, while mastectomy with breast reconstruction is an alternative for those who are not eligible for Breast-conserving surgery. Several studies have compared the quality of life and patient satisfaction among individuals receiving different types of surgery (Breast-conserving surgery, mastectomy alone, or mastectomy with reconstruction). For example, Meghan R. demonstrated that patients undergoing Breast-conserving surgery experience a higher quality of life compared to those undergoing mastectomy with breast reconstruction, whereas J. Dauplat's study showed that patients who undergo mastectomy with breast reconstruction report a higher quality of life than those who undergo mastectomy alone.

However, the investigators hypothesize that the advantages of a specific type of surgery over another, such as Breast-conserving surgery versus breast reconstruction, may vary among patients with different socioeconomic factors. For instance, the benefits of breast reconstruction over Breast-conserving surgery might be more pronounced in young patients who require a more socially active lifestyle.

Additionally, the benefits of one type of surgery over another may also vary at different time points during post-operative follow-up. Furthermore, it is worth noting that most current studies have been conducted in Caucasian populations. In contrast to Caucasians, Asians typically have smaller breast volumes, potentially leading to more significant defects after Breast-conserving surgery and possibly poorer aesthetic outcomes. Therefore, a study focusing on Asian young breast cancer populations is necessary.

DETAILED DESCRIPTION:
This study is a prospective, observational cohort study aiming to enroll 1000 young Chinese breast cancer patients and assign them to three arms: Breast-conserving surgery, mastectomy alone, and mastectomy with breast reconstruction, based on their clinical decisions and preferences. Clinicopathological features (age,Tumor, Node, Metastasis stages, pathological features, etc.), socioeconomic determinants (education level, income, insurance status, marital status, occupational status, personality, etc.), treatment information (neoadjuvant chemotherapy or not, post-operative complications), and survival (local recurrence, metastasis) will be recorded.

All patients will be followed at 6 and 12 months for the first year after diagnosis, then yearly thereafter for an additional 9 years (for a total follow-up of at least 10 years following diagnosis). During the post-operative follow-up, quality of life, psychological well-being, decision regret, surgical information, treatment costs, and surveillance-follow-up will be recorded.

The primary endpoint of this study is the quality of life, assessed using the Breast-Q and the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Secondary endpoints include decisional conflict scale, decision regret scales, and the Hospital Anxiety and Depression Scale (HADS).

The primary and secondary endpoints will be compared among the three arms, and the impact of socioeconomic determinants at baseline on these endpoints will also be investigated. Additionally, the investigators aim to explore the potential of a novel subtyping method for young breast cancer patients using selected socioeconomic determinants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old.
* The surgery time and procedure have been confirmed, and the surgical informed consent and research informed consent forms have been signed.
* Informed consent obtained from patient.
* Unilateral Breast Cancer.
* Good health,the patient is able to tolerate general anesthesia and surgery, with an ECOG performance status of ≤2 points.
* No history of breast/axillary radiation therapy.
* Willing and capable of complying with the study protocol visits, treatment plans, and other research procedures.

Exclusion Criteria:

* Bilateral breast cancer.
* Inflammatory breast cancer.
* Stage IV breast cancer.
* Physical examination and imaging suggest tumor infiltration into the skin, pectoralis major muscle, and other adjacent tissues.
* Patients unable to tolerate surgery due to coagulation abnormalities.
* In patients without evidence of breast cancer in the contralateral breast, requesting contralateral prophylactic mastectomy.
* In patients who have undergone surgical treatment for breast cancer (including mastectomy, breast-conserving surgery, and mastectomy with implant reconstruction), requesting secondary breast surgery.
* Patients with a history or current diagnosis of other malignancies, excluding thyroid cancer.
* The conditions considered unsuitable for inclusion by researchers.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Young breast cancer women.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2035-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Participant's breast satisfaction assessed by BREAST-Q questionnaire version 2.0 | Pre-operation and 10 years
  Utilizing the BREAST-Q questionnaire, this measure assesses women's self-reported satisfaction with their breasts and associated quality of life, encompassing psychosocial, sexual, and physical well-being. Scores range from 0 (worst) to 100 (best), with higher scores indicating a more favorable outcome.Assessment is conducted preoperatively and 10 years postoperatively.
Participant's health-related quality of life assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | 10 years
  Assessed through the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), this self-administered questionnaire consists of 30 items designed to evaluate the health-related quality of life among cancer patients. For questions 1 to 28, a 4-point scale is used, ranging from 1 ("Not at all") to 4 ("Very much"), with lower scores indicating a more positive outcome. Questions 29 and 30 employ a 7-point scale, with scores ranging from 1 ("Very poor") to 7 ("Excellent"), where higher scores signify a better outcome.Assessment is conducted 10 years postoperatively.

SECONDARY OUTCOMES:
Participant's decisional conflict assessed by Decisional Conflict Scale questionnaire | Pre-Operative
  Administered pre-operation, this tool evaluates the patient's conflict regarding the decision for surgery. Each item is rated on a Likert Scale with five responses, ranging from 0 ("Not at All") to 4 ("Extremely"), resulting in a total score ranging from 0 (Less conflicted) to 100 (Highly conflicted).Assessment is conducted preoperatively.
Participant's decision regret assessed by Decision Regret Scale questionnaire | 10 years
  Conducted during follow-up sessions, this assessment captures the patient's sentiments and remorse regarding the treatment-related decision to undergo surgery. Five items specifically inquire about feelings of regret. Scores range from 0 to 100, with a higher score indicating a greater level of decision-related regret.Assessment is conducted 10 years postoperatively.
Participant's anxiety and depression assessed by Hospital Anxiety and Depression Scale questionnaire | Pre-operation and 10 years
  Administered during follow-ups, this scale measures the patient's psychological change. The HADS comprises two 7-item subscales assessing depression and anxiety symptoms separately. Higher scores indicate greater levels of depression and/or anxiety.Assessment is conducted preoperatively and 10 years postoperatively.

OTHER OUTCOMES:
Influence of Socioeconomic, Psychological, and Clinicopathological Factors on Outcomes | Pre-operation and 10 years
  Exploring the Influence of Socioeconomic, Psychological, and Clinicopathological Features on Primary and Secondary Outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The study protocol and the raw and clean data for analysis will be shared among the participated researchers. Non-researchers could obtain relevant informations from the researchers upon reasonable requests.

REFERENCES:
- [Background] Dominici L, Hu J, Zheng Y, Kim HJ, King TA, Ruddy KJ, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Warner E, Wong JS, Partridge AH, Rosenberg SM. Association of Local Therapy With Quality-of-Life Outcomes in Young Women With Breast Cancer. JAMA Surg. 2021 Oct 1;156(10):e213758. doi: 10.1001/jamasurg.2021.3758. Epub 2021 Oct 13. PMID 34468718
- [Background] Hanson SE, Lei X, Roubaud MS, DeSnyder SM, Caudle AS, Shaitelman SF, Hoffman KE, Smith GL, Jagsi R, Peterson SK, Smith BD. Long-term Quality of Life in Patients With Breast Cancer After Breast Conservation vs Mastectomy and Reconstruction. JAMA Surg. 2022 Jun 1;157(6):e220631. doi: 10.1001/jamasurg.2022.0631. Epub 2022 Jun 8. PMID 35416926
- [Background] Diao K, Lei X, He W, Jagsi R, Giordano SH, Smith GL, Caudle A, Shen Y, Peterson SK, Smith BD. Patient-reported Quality of Life After Breast-conserving Surgery With Radiotherapy Versus Mastectomy and Reconstruction. Ann Surg. 2023 Nov 1;278(5):e1096-e1102. doi: 10.1097/SLA.0000000000005920. Epub 2023 May 26. PMID 37232937
- [Background] Rosenberg SM, Dominici LS, Gelber S, Poorvu PD, Ruddy KJ, Wong JS, Tamimi RM, Schapira L, Come S, Peppercorn JM, Borges VF, Partridge AH. Association of Breast Cancer Surgery With Quality of Life and Psychosocial Well-being in Young Breast Cancer Survivors. JAMA Surg. 2020 Nov 1;155(11):1035-1042. doi: 10.1001/jamasurg.2020.3325. PMID 32936216
- [Background] Riba LA, Gruner RA, Alapati A, James TA. Association between socioeconomic factors and outcomes in breast cancer. Breast J. 2019 May;25(3):488-492. doi: 10.1111/tbj.13250. Epub 2019 Apr 15. PMID 30983100
- [Background] Flanagan MR, Zabor EC, Romanoff A, Fuzesi S, Stempel M, Mehrara BJ, Morrow M, Pusic AL, Gemignani ML. A Comparison of Patient-Reported Outcomes After Breast-Conserving Surgery and Mastectomy with Implant Breast Reconstruction. Ann Surg Oncol. 2019 Oct;26(10):3133-3140. doi: 10.1245/s10434-019-07548-9. Epub 2019 Jul 24. PMID 31342397
- [Background] Dauplat J, Kwiatkowski F, Rouanet P, Delay E, Clough K, Verhaeghe JL, Raoust I, Houvenaeghel G, Lemasurier P, Thivat E, Pomel C; STIC-RMI working group. Quality of life after mastectomy with or without immediate breast reconstruction. Br J Surg. 2017 Aug;104(9):1197-1206. doi: 10.1002/bjs.10537. Epub 2017 Apr 12. PMID 28401542